CLINICAL TRIAL: NCT03108209
Title: Evaluation of the Interest and Tolerance of a Photoprotection Strategy in Prevention of Phototoxicities in Patients Undergoing Vemurafenib Treatment Associated or Not With Cobimetinib
Brief Title: Prevention of Phototoxicities in Patients Undergoing Vemurafenib Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michele Sayag (Industry)
Responsible Party: Sponsor-Investigator, Michele Sayag, Dr, NAOS Institute of Life Science
Organization: NAOS Institute of Life Science (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RC2015/PhMZb/Fr/TCO04915
Record Dates: First submitted 2017-03-14; First posted 2017-04-11 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Phototoxicity
MeSH Terms: conditions — Dermatitis, Phototoxic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm (Experimental): Signle arm study. Every subjects apply Photoderm Max lait SPF50+ and Photoderm stick SPF50+
  Interventions: Other: Photoderm Max lait SPF50+; Other: Photoderm Max Stick SPF50+

INTERVENTIONS:
Other: Photoderm Max lait SPF50+ — Subjects apply Photoderm Max lait SPF50+ at the beginning of their treatment by Vemurafenib/Cobimetinib in prevention of phototoxicities
Other: Photoderm Max Stick SPF50+ — Subjects apply Photoderm Max Stick SPF50+ at the beginning of their treatment by Vemurafenib/Cobimetinib in prevention of phototoxicities

SUMMARY:
Vemurafenib is an anti-cancer treatment indicated as monotherapy in the treatment of adult patients with non-resectable or metastatic melanoma carrying a BRAF V600 mutation.

Cobimetinib is indicated in combination with Vemurafenib in the treatment of adult patients with non-resectable or metastatic melanoma carrying a BRAF V600 mutation.

These treatments are associated with a lot of adverse reactions, which may lead to dose reduction, temporary interruption or discontinuation of treatment, which often leads to treatment failure or a decrease in treatment compliance.

The most commonly reported adverse reactions (> 30%) with Vemurafenib are arthralgia, rash, photosensitivity reaction, nausea, alopecia and pruritus. The most commonly reported adverse events (> 20%) associated with Cobimetinib / Vemurafenib are diarrhea, rash, nausea, pyrexia, photosensitivity reaction, increase of alanine aminotransferase, elevation of aspartate aminotransferase, blood creatine phosphokinase elevation and vomiting.

The risk of presenting a phototoxicity adverse event with Vemurafenib in monotherapy or in combination with Cobimetinib is very common (≥ 1/10) according to MedDRA.

The use of optimal photoprotection including the repeated daily use of external photoprotection products is currently recommended for all patients receiving treatment with vemurafenib or with the combination of vemurafenib and cobimetinib.

DETAILED DESCRIPTION:
Vemurafenib is an anti-cancer treatment indicated as monotherapy in the treatment of adult patients with non-resectable or metastatic melanoma carrying a BRAF V600 mutation.

Cobimetinib is indicated in combination with Vemurafenib in the treatment of adult patients with non-resectable or metastatic melanoma carrying a BRAF V600 mutation.

These treatments are associated with a lot of adverse reactions, which may lead to dose reduction, temporary interruption or discontinuation of treatment, which often leads to treatment failure or a decrease in treatment compliance.

The most commonly reported adverse reactions (> 30%) with Vemurafenib are arthralgia, rash, photosensitivity reaction, nausea, alopecia and pruritus. The most commonly reported adverse events (> 20%) associated with Cobimetinib / Vemurafenib are diarrhea, rash, nausea, pyrexia, photosensitivity reaction, increase of alanine aminotransferase, elevation of aspartate aminotransferase, blood creatine phosphokinase elevation and vomiting.

The risk of presenting a phototoxicity adverse event with Vemurafenib in monotherapy or in combination with Cobimetinib is very common (≥ 1/10) according to MedDRA.

Two studies on Vemurafenib as monotherapy have demonstrated these results. One study concerns 468 patients from a randomized, open-label Phase III study in adult patients with non-resectable melanoma or stage IV with a BRAF V600 mutation, the other is a study Phase II study in a single group of patients with stage IV melanoma carrying a BRAF V600 mutation after failure of at least one prior systemic treatment. The study on the combination of Vemurafenib and Cobimetinib is a randomized, double-blind, placebo-controlled phase III study (GO28141), which evaluated Cobimetinib in combination with vemurafenib compared to vemurafenib alone Of patients with non-resectable (stage III) or metastatic (stage IV) melanoma carrying a BRAF V600 mutation naive from any treatment.

The use of optimal photoprotection including the repeated daily use of external photoprotection products is currently recommended for all patients receiving treatment with vemurafenib or with the combination of vemurafenib and cobimetinib.

The objective of the study is to demonstrate that the application of Photoderm Max SPF50 + Milk (UVA / UVB broad spectrum sunscreen) associated with the application of the Photoderm Max SPF50 + stick (SPF ≥ 50) on the first day of treatment with Vemurafenib or its combination with cobimetinib reduces the occurrence of this adverse event from a frequency (≥ 1/10) to a frequency (≤ 1/10) with regular application to all exposed areas.

ELIGIBILITY:
Inclusion Criteria:

* Subject naive of i-BRAF treatment, receiving a Vemurafenib treatment in association or not with Cobimetinib in 1st or 2nd line of treatment in non resecable metastatic melonoma with BRAF V600 mutation;
* Subject aged 18 or older ;
* Subject who can be follow regularly by the investigator ;
* Informed and consent subjects who read and signed the ICF ;
* Subject who does not participate in another study, exepted therapeutic clinical trial with Vemurafenib in association or not with Cobimetinib ;
* Compliant subject, left to the discretion of the investigator.

Exclusion Criteria:

* Pregnant or lactating women
* Women of reproductive age without contraception deemed effective for at least 1 month
* For women of reproductive age receiving Cobimetinib treatment, lack of use of two effective methods of contraception, such as a condom or other barrier method (with spermicide if available).
* Subject having a history of allergy to an ingredient of the tested products
* Subject with skin sensitivity to sunscreens or any of the components of the products under investigation
* Subjects taking another photosensitising treatment (left to the discretion of the investigator)
* Subject presenting a concomitant pathology which may interfere with the course of the study (left to the discretion of the investigator)
* Subjects with cutaneous photosensitivity or systemic disease including: lupus, dermatomyositis, porphyria, lucite ... (non-exhaustive list left to the discretion of the investigator).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-07; Primary Completion 2017-12 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Number of photosensitivity reactions as assessed by CTCAE v4.03 | 3 months
  Decrease of photosensitivity reaction frequency (in total number of reaction) compared to what is described in the Summary of Product Characteristics of Vemurafenib (photosensitivity reactions are described as very common ≥ 1/10)

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte Dreno, MD, Principal Investigator — Nantes University Hospital
Locations (1):
- CHU Nantes, Nantes, France

IPD SHARING:
Plan to Share IPD: No